CLINICAL TRIAL: NCT06998797
Title: Efficacy of Subcutaneous Infliximab in Acute Severe Ulcerative Colitis: a Multicenter Retrospective Study
Acronym: ISAC
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, CARON Bénédicte, MD, PhD, Central Hospital, Nancy, France
Other Study IDs: 2025PI032
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Global cohort
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data collection from medical records

SUMMARY:
Around 25% of patients with ulcerative colitis will develop acute severe colitis during the course of their disease. The first-line treatment for acute severe colitis is intravenous corticosteroid therapy. In case of a cortico-resistant form, treatment with intravenous (ciclosporin or Infliximab is indicated), according to European guidelines.

The emergence of biosimilar in the last years is a turning point in a context of optimizing healthcare costs and improving patient quality of life, with the arrival of the subcutaneous form of Infliximab in 2020, with similar results in terms of clinical remission, but also blood levels of Infliximab compared with the intravenous form. To our knowledge, there are very few data on the use of subcutaneous Infliximab after intravenous induction in patients with acute severe colitis.

The aim of this study is to evaluate the efficacy of subcutaneous Infliximab in ulcerative colitis patients with acute severe colitis, and the factors associated with treatment failure.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old
* Diagnosis of acute severe ulcerative colitis according to Truelove Witts criteria
* Patients treated with at least one injection of subcutaneous Infliximab after induction with two or three intravenous perfusions of Infliximab
* Patients with a follow-up of at least 12 months after the first subcutaneous injection
* 12-month data available in medical records
* Patient who has received full information about the organization of the research and who has not objected to his or her participation and to the use of his or her data.

Exclusion Criteria:

* Patients with intravenous Infliximab as a maintenance treatment
* Patients switched from intravenous to subcutaneous form during follow-up, and who received more than three intravenous perfusions
* Protected persons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in acute severe ulcerative colitis treated with subcutaneous Infliximab
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Treatment failure at 12 months to describe treatment effectiveness | After study completion, average of 1 month
  Absence of steroid free clinical remission (Mayo score ≤2, with every sub-score ≤1) or absence of endoscopic response (Mayo endoscopic sub-score ≤1) or use of a rescue treatment if relapse (other than Infliximab) or occurrence of a severe adverse event with withdrawal of treatment or colectomy or death during follow-up

IPD SHARING:
Plan to Share IPD: Undecided